CLINICAL TRIAL: NCT01186887
Title: A Trial Assessing the Outcome of Celecoxib Administration Versus Placebo Following Anterior Cruciate Ligament Reconstruction
Brief Title: A Trial Assessing the Outcome of Celecoxib Administration Versus Placebo Following Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-645
Record Dates: First submitted 2010-03-17; First posted 2010-08-23 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: primary ACL reconstruction with a hamstring graft
MeSH Terms: conditions — Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib (Placebo Comparator)
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — The treatment group will receive 400 mg Celecoxib p.o. preoperatively and the control group will receive a placebo between 1 and 3 hours pre-op, when other standard medications are administered. The treatment group will receive 200 mg of Celecoxib orally twice per day post operatively, for a duration of 5 days based on dosing protocols shown to be well tolerated and effective in treating pain following ambulatory surgery. The control group will receive a 5 day supply of placebo pills. Both groups will receive standard post surgical narcotic prescription (Oxycodone IR 5 - 10 mg po qid prn and acetaminophen 325 - 650 mg PO qid prn
  Arms: Celecoxib
Drug: Placebo — The treatment group will receive 400 mg Celecoxib p.o. preoperatively and the control group will receive a placebo between 1 and 3 hours pre-op, when other standard medications are administered. The treatment group will receive 200 mg of Celecoxib orally twice per day post operatively, for a duration of 5 days based on dosing protocols shown to be well tolerated and effective in treating pain following ambulatory surgery. The control group will receive a 5 day supply of placebo pills. Both groups will receive standard post surgical narcotic prescription (Oxycodone IR 5 - 10 mg po qid prn and acetaminophen 325 - 650 mg PO qid prn
  Arms: Placebo

SUMMARY:
The aim of this study is to directly compare the clinical outcomes of both the celecoxib and placebo groups following anterior cruciate ligament (ACL) reconstruction. The study will have short and long term goals. Validated outcome measures will aim to quantify pain control at 2 weeks after surgery, as well as knee function at 2 year follow-up. Groups will be compared using pain control scales, and functional knee outcome scores. The first null hypothesis tested by this study is that the celecoxib group experiences equal pain control compared with the placebo group. The second null hypothesis is that no knee function difference will be found between the celecoxib and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Any patient 18 years and over undergoing primary anterior cruciate ligament reconstruction with hamstring grafts will be considered for this study.

Exclusion Criteria:

* Patients will be excluded if they have bilateral ACL injuries, require revision ACL reconstruction, require meniscus repair, have multiple ligament injuries, gross osteoarthritis, significant clinical malalignment or if they cannot attend appropriate follow-up. Other exclusion criteria will include use of a regional block during the surgery, a diagnosis of esophageal, gastric, or duodenal ulceration, hepatic disease, renal disease, hypertension, hypersensitivity to Celecoxib, known allergic-type reactions to sulfonamides, known allergies to ASA or other NSAIDS, inflammatory bowel disease or hyperkalemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to test the null hypothesis that Celecoxib perioperatively does not negatively influence the static testing of ACL reconstruction as measured by KT arthrometer at 2 years post op. | 2 years

SECONDARY OUTCOMES:
The 2nd outcome tested by this study is that the celecoxib group experiences equal pain control compared with the placebo group. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Dervin, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada